CLINICAL TRIAL: NCT04582409
Title: A Randomized, Placebo-controlled, Investigator- and Participant-blinded Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of HSY244 in Participants With Atrial Fibrillation
Brief Title: A Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of HSY244 in Participants With Atrial Fibrillation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to business decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHSY244X2201; 2020-004327-17 (EudraCT Number)
Record Dates: First submitted 2020-10-07; First posted 2020-10-09 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; arrhythmia; pharmacological cardioversion
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HSY244 (Experimental): HSY244 150 mg concentrate solution for injection via intravenous infusion
  Interventions: Drug: HSY244
- Placebo (Placebo Comparator): Placebo concentrate solution for injection via intravenous infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HSY244 — HSY244 concentrate solution for injection via intravenous infusion
  Arms: HSY244
Other: Placebo — Placebo concentrate solution for injection via intravenous infusion
  Arms: Placebo

SUMMARY:
This was a randomized, placebo-controlled, investigator- and participant-blinded study to evaluate the efficacy, safety, tolerability, and pharmacokinetics (PK) of HSY244 in participants with atrial fibrillation (AF), with and without heart failure (HF).

DETAILED DESCRIPTION:
A screening period of up to 3 days (72 hours) was used to assess eligibility. After eligibility was confirmed, patients were randomized to either HSY244 or placebo. Prior to study drug administration, pre-dose assessments were completed. After the start of study drug administration, the participant was monitored for cardioversion to sinus rhythm. If a participant was still in AF at 90 minutes after the start of study drug administration, direct current cardioversion was planned to be applied at a time deemed appropriate by the investigator.

ELIGIBILITY:
Key Inclusion Criteria:

* At screening, written informed consent were required to be obtained before any assessment was performed and only participants able to provide written informed consent themselves were included in this study.
* Hemodynamically stable men and women (either of non-child-bearing potential or child bearing potential with highly effective contraception) between 18 and 80 years of age (inclusive) at screening with a clinical indication for direct current cardioversion of AF.
* At screening, current episode of AF had been ongoing for ≥6 hours and ≤60 days
* Successful initiation and achievement of therapeutic levels of national guideline and institution-specific anticoagulation therapy as appropriate for the duration of the AF episode and risk for the participant.
* Completion of national guideline and institution-specific imaging evaluation for left atrial thrombi as appropriate for the duration of AF episode and risk for the participant.
* At screening, participants were required to weigh at least 60 kg to participate in the study and were required to have a body mass index (BMI) within the range of 18 - 45 kg/m^2. BMI = Body weight (kg) / [Height (m)]^2
* At screening, vital signs (systolic blood pressure and pulse rate) were assessed in the sitting position. Sitting vital signs were required to be within the following ranges (exclusive):

  * systolic blood pressure between 100-160 mmHg and diastolic blood pressure 60-100 mmHg
  * pulse rate (ventricular rate) between 60-120 bpm.

Key Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they were using highly effective methods of contraception during dosing and for 4 days after stopping of investigational drug.
* Sexually active males unwilling to use a condom during intercourse while taking investigational drug and for 96 hours after study drug administration. A condom was required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of the investigational drug via seminal fluid to their partner. In addition, male participants could not donate sperm for the time period specified above.
* Use of any anti-arrhythmic class I or III drug (including Ranolazine [Ranexa]) within 5 half lives before randomization; including use of amiodarone within 3 months before randomization.
* At screening, history of current diagnosis of ECG abnormalities or cardiac rhythm disorders as determined by the Investigator's interpretation of the ECG findings indicating a significant risk for participating in the study, such as:

  * History of Torsades de Pointes (TdP), any other polymorphic ventricular tachycardia, sustained monomorphic ventricular tachycardia, long QT syndrome, or Brugada syndrome.
  * Wolfe-Parkinson-White (WPW) syndrome
  * In the absence of a complete bundle branch block a resting QTcF >460 msec for men and >470 msec for women (mean of ≥ 5 consecutive QT intervals)
  * In the presence of a complete bundle branch block, a prolonged QTcF or JTc that, in the opinion of the investigator, may pose a risk to patient safety
  * Third-degree (complete) heart block, or second-degree Mobitz type II heart block
* Attempted or unsuccessful cardioversion within 2 weeks prior to randomization.
* Presence of known severe mitral regurgitation and/or known severely dilated left atrium.
* Pre-existing or tachycardia-induced moderate to severe cardiac dysfunction (New York Heart Association Class III and IV).
* History within the preceding 3 months prior to randomization of: myocardial infarction, unstable angina, cardiac surgery, or a percutaneous coronary intervention.
* History of a confirmed stroke or transient ischemic attack (TIA).
* History or current diagnosis of any seizure disorder, epilepsy, significant head trauma, or other disorders increasing the risk for seizures.
* History or current diagnosis of a major neurologic or psychiatric disorder that, in the opinion of the investigator, poses a risk to patient safety to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (2):
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Lansing, Michigan
- Germany (2):
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Frankfurt

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: Results for CHSY244X2201 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18069
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1719

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A screening period of up to 3 days (72 hours) was used to assess eligibility.
Period: Overall Study
Arm/Group | HSY244 | Placebo
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HSY244 | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.73) | 60.0 (4.05) | 60.3 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 6 | 6 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 5 | 12
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Conversion to Sinus Rhythm for at Least 1 Minute Within 90 Minutes From the Start of Study Drug Administration.
Description: Conversion to sinus rhythm was monitored using a Holter monitoring device through 90 minutes after the start of study drug administration.
  If a participant had been monitored for at least 45 minutes and did not convert to sinus rhythm for at least one minute, the primary endpoint was defined as 'no'. If a participant converted to sinus rhythm for at least one minute at any time during the post-treatment 90 minutes observation period, regardless of the length of time monitored, the primary endpoint was to be defined as 'yes'.
Time Frame: 90 minutes from the start of study drug administration
Population: Pharmacodynamic (PD) analysis set: Participants with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Count of Participants; unit: Participants
Arm/Group | HSY244 | Placebo
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The Cmax is the maximum (peak) observed plasma drug concentration after single-dose administration.
  Actual recorded sampling times were taken into consideration for PK calculations.
Time Frame: Day 1 (0 min (pre-dose), 15 min (end of infusion), 30 min , 60 min, 90 min and 180 min) and Day 5
Population: Pharmacokinetic (PK) analysis set: Participants with at least one available valid PK concentration measurement, who received the investigational product and with no protocol deviations that impact on PK data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HSY244 | Placebo
Number analyzed (Participants) | 7 | 0
ng/mL | 4800 (3890) |

3. Secondary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Description: Tmax is the time to reach maximum (peak) plasma drug concentration after single dose administration (time).
  Actual recorded sampling times were taken into consideration for PK calculations.
Time Frame: Day 1 (0 min (pre-dose), 15 min (end of infusion), 30 min , 60 min, 90 min and 180 min) and Day 5
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour
Arm/Group | HSY244 | Placebo
Number analyzed (Participants) | 7 | 0
Hour | 0.28 [0.25 to 0.30] |

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUClast)
Description: AUClast is the AUC from time zero to the last measurable concentration sampling time (tlast).
  Actual recorded sampling times were taken into consideration for PK calculations.
Time Frame: Day 1 (0 min (pre-dose), 15 min (end of infusion), 30 min , 60 min, 90 min and 180 min) and Day 5
Population: Pharmacokinetic (PK) analysis set: Participants with at least one available valid PK concentration measurement, who received the investigational product and with no protocol deviations that impact on PK data. Only participants with available AUClast data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | HSY244 | Placebo
Number analyzed (Participants) | 6 | 0
h*ng/mL | 2960 (1510) |

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 31 days.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up
Groups:
- Total: Total
Arm/Group | HSY244 | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/6 | 1/13
Other Adverse Events (participants affected / at risk) | 6/7 | 5/6 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HSY244 (N=7) | Placebo (N=6) | Total (N=13)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HSY244 (N=7) | Placebo (N=6) | Total (N=13)
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Infusion site pain (General disorders) | 0 | 1 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood pressure increased (Investigations) | 2 | 0 | 2
Blood urine present (Investigations) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT04582409/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT04582409/SAP_001.pdf